CLINICAL TRIAL: NCT05516537
Title: Promotion of Exercise Behavior Among Rural-Residing African-Americans With Multiple Sclerosis
Brief Title: Examining the Effects of a Remotely-delivered, Racially-tailored Exercise Training Program for Immediate and Sustained Improvements in Walking Dysfunction, Symptoms, and Health-related Quality of Life (HRQOL) Among African-Americans With Multiple Sclerosis (MS) Residing in Rural Environments.
Acronym: TEAAMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Alabama at Birmingham (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Robert W Motl, Robert W. Motl, PhD, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0526; 20016 (Other Grant/Funding Number: Bristol Myers Squibb Foundation)
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: Rural; Walking dysfunction; Health-Related Quality of Life; African-American
MeSH Terms: conditions — Multiple Sclerosis | interventions — Guidelines as Topic; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guidelines for Exercise in Multiple Sclerosis (GEMS) (Experimental): Participants in this condition will receive a 4-month home-based, remotely supported aerobic and resistance exercise program based on the Guidelines for Exercise in Multiple Sclerosis (GEMS).
  Interventions: Behavioral: Guidelines for Exercise in Multiple Sclerosis (GEMS)
- FLEX Stretching and Toning Program (Sham Comparator): Participants in this condition will receive a 4-month home-based, remotely supported stretching program emphasizing flexibility and range of motion as important components of fitness based on Stretching for People with MS: An Illustrated Manual from the National MS Society.
  Interventions: Behavioral: FLEX Stretching and Toning Program

INTERVENTIONS:
Behavioral: Guidelines for Exercise in Multiple Sclerosis (GEMS) — Remotely-coached/guided, home-based program delivered using telerehabilitation focusing on aerobic fitness and muscle strength as a mode of training.
  Arms: Guidelines for Exercise in Multiple Sclerosis (GEMS)
Behavioral: FLEX Stretching and Toning Program — Remotely-coached/guided, home-based program delivered using telerehabilitation focusing on stretching and range of motion as the mode of training.
  Arms: FLEX Stretching and Toning Program

SUMMARY:
The proposed project involves a high-quality randomized controlled (RCT) design that examines the effects of a remotely-delivered, racially-tailored exercise training program for immediate and sustained improvement in walking dysfunction, symptoms, and health-related quality of life (HRQOL) among African-Americans with MS residing in rural environments. The primary analysis will test the hypothesis that those who are randomly assigned into the intervention condition (i.e., exercise training) will demonstrate (a) improvements in outcomes from baseline that (b) are sustained over 4-months of follow-up compared with those in the control condition (i.e., stretching).

DETAILED DESCRIPTION:
There is a lack of evidence from high-quality randomized controlled trials (RCTs) of exercise training for African-Americans with multiple sclerosis (MS), as only 1.7% of participants in physical activity and exercise research involving persons with MS identify as African-American. The population of African-Americans with MS deserves equal and focal research that addresses the unique challenges of MS in the African-American rural residing community. We uniquely address this population with a highly-developed and refined exercise training program that is racially-tailored for the target population. We further provide a highly-developed and refined exercise training program that can be undertaken in one's home and/or local community, and does not require facility access that is extremely limited in the target, rural residing population of persons with MS. The program is further tailored based on qualitative research and addresses the unique needs of the African-American community with MS. There is no other research program this advanced in study refinement and design for immediate integration into a high-quality RCT for changing the lives of African-Americans with MS who reside in rural communities of the Southeastern portion of the United States. If successful, the study, as designed, will provide Class I evidence that is necessary for immediate implementation after trial completion through insurance providers and healthcare providers, including physical therapists, rehabilitation practitioners, and community health workers/providers. This program further aligns with recently developed and highly-refined conceptual and practice models for implementation of exercise into the care of persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* English as primary language
* Identify as African-American or Black
* Age of 18 years or older
* Diagnosis of MS
* Relapse free in the past 30 days
* Internet and email access
* Willingness to complete the outcome questionnaires
* Willingness to undergo randomization
* Insufficient physical activity (not meeting current physical activity guidelines based on GLTEQ)
* Mild-moderate ambulatory disability (MSWS-12 score between 25-49 & PDDS score between 2-4)

Exclusion Criteria:

* Individuals not meeting above inclusion criteria
* Individuals with moderate to high risk for contraindications of possible injury or death when undertaking strenuous or maximal exercise (PARQ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Walking Dysfunction | Changes in walking scores from Baseline, 4-months, and 8-months.
  Multiple Sclerosis Walking Scale-12 (MSWS-12); scores range between 0 (min) and 100 (max), higher scores reflect greater walking problems.

SECONDARY OUTCOMES:
Disability | Changes in disability scores from Baseline, 4-months, and 8 months.
  Patient Determined Disease Steps (PDDS) scale; scores range between 0 (min) and 8 (max), higher score reflect greater perceived disability.
Fatigue Severity | Changes in fatigue from Baseline, after 4-month intervention period, and 4 months after intervention cessation.
  Fatigue Severity Scale (FSS); scores range between 1 (min) and 7 (max), higher scores reflect greater fatigue severity.
Depressive Symptoms | Changes in depressive symptoms from Baseline, after 4-month intervention period, and 4 months after intervention cessation.
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms.
Anxiety | Changes in anxiety symptoms from Baseline, after 4-month intervention period, and 4 months after intervention cessation.
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms.
Health-related Quality of Life (HRQOL) | Changes in quality of life from Baseline, after 4-month intervention period, and 4 months after intervention cessation.
  Multiple Sclerosis Impact Scale (MSIS-29); scores range between 0 (min) and 100 (max), higher scores indicate greater impact of disease on daily function (i.e. worse outcomes).

OTHER OUTCOMES:
Exercise Behavior | Changes in exercise behavior from Baseline, after 4-month intervention period, and 4 months after intervention cessation.
  Godin Leisure Time Exercise Questionnaire (GLTEQ); scores range between 0 (min) and 119 (max), higher scores indicate greater engagement in exercise behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Motl, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No